CLINICAL TRIAL: NCT05914441
Title: Development Of Spanish-Portuguese Thrombotic Thrombocytopenic Purpura Registry (REPTT): A Study Proposal Of The Spanish Society Of Hematology And Hemotherapy (SEHH) Whit The Portuguese Society Of Hematology (SPH)
Brief Title: Spanish-Portuguese Thrombotic Thrombocytopenic Purpura Registry
Acronym: RE-PTT
Status: Recruiting | Type: Observational
Sponsor: Fundación Española de Hematología y Hemoterapía (Other)
Responsible Party: Sponsor
Other Study IDs: RE-PTT
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Purpura, Thrombocytopenic
Keywords: registry; Thrombotic thrombocytopenic purpura; real-world; observational
MeSH Terms: conditions — Purpura, Thrombocytopenic; Purpura, Thrombotic Thrombocytopenic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — This project will be linked to obtaining biological samples for a serum and DNA library from patients with TTP, to study the impact of the molecular / biological factors on the short and long-term prognosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thrombotic thrombocytopenic purpura patients: Including all patients enrolled in the study
  Interventions: Other: Standard clinical practice

INTERVENTIONS:
Other: Standard clinical practice — The study will be carried out in the context of the usual clinical practice conditions, not imposing restrictions on the participating physician or influencing their normal clinical practice.

SUMMARY:
REPTT is an observational, prospective, multi-country, multicentre and non-interventional registry in which at least 300 patients with Thrombotic thrombocytopenic purpura (TTP) in Spain and Portugal will be evaluated.

The study will be carried out in the context of the usual clinical practice conditions, not imposing restrictions on the participating physician or influencing their normal clinical practice.

DETAILED DESCRIPTION:
TTP is a rare life-threatening haematological disease characterised by thrombotic microangiopathy (TMA) with an average annual prevalence of approximately 10 cases/million people worldwide and an annual incidence between 1.5 and 6.0 cases per million according to different studies conducted in France, the United States and in the United Kingdom. In Spain the incidence is 2,67 cases / million population per year.

Acute TTP episodes cause sequelae like vascular disease or kidney damage along with other symptoms more subtle like small neurocognitive deficits and myocardial infarction.

Thus, prompt resolution of acute episodes along with a better understanding of the cardiac abnormalities may allow to prevent further complications, to develop targeted rehabilitation techniques for TTP patients and to improve their quality of life.

This project will collect a big database capable of providing better answers to questions related with treatment efficacy, associated morbidity and mortality, and the possible neurocognitive and cardiac sequelae derived from relapses and acute episodes. Additionally, this project will be linked to obtaining biological samples for a serum and DNA library from patients with TTP.

Patients will be recruited by medical researchers specialized in haematology or by other investigators specialized in thrombotic microangiopathies disease management. This recruitment will be performed in a competitive manner. The collection period will be at least 3 years with the possibility of extending it.

REPTT aims to evaluate new scores and prognostic factors of morbidity and mortality in TTP patients.

The final aim is to establish guidelines and recommendation to improve the global management, diagnosis and treatment of patients with TTP in real-life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diagnosis of TTP according to International Consensus criteria from centres in Spain and Portugal.
2. Patients that voluntarily sign the informed consent. For subjects unable to provide informed consent, a fully recognized medical authority may be used according to local laws.
3. Patients between 0 to 99 years old at the time of diagnosis.

Note: Decision was taken to treat the patient with an specific treatment prior and independently of patient inclusion in this non interventional study.

Exclusion Criteria:

1. Inability to comply with study procedures and follow-up exams.
2. Patients with any type of alteration that compromises their ability to grant written informed consent.
3. Patients that do not consent to participate in the study and do not sign informed consent.
4. Patients that do not meet the criteria previously mentioned for TTP.

Max Age: 99 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with Thrombotic thrombocytopenic purpura (TTP)
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of TTP in Spain/Portugal | Throughout the study period, calculated for the 3 years of expected duration.
  Number of patients diagnosed with TTP and enrolled in the registry per year
Morbidity of TTP in Spain/Portugal | Throughout the study period, calculated for the 3 years of expected duration.
  Percentage of patients diagnosed with TTP and enrolled in the registry among spanish / portuguese population per year
Mortality of TTP in Spain/Portugal | Throughout the study period, calculated for the 3 years of expected duration.
  Percentage of patients diagnosed with TTP and enrolled in the registry per year who died due to the disease

SECONDARY OUTCOMES:
Clinical response to treatment rate | Throughout the study period, approximately 3 years per patient
  Defined as sustained normalization of platelet counts above the lower limit of the established reference range and of lactate dehydrogenase (LDH) after cessation of plasma exchange. The number of patients that achieved clinical response and their frequency will be reported.
TTP Clinical remission rate | Throughout the study period, approximately 3 years per patient
  Defined as a clinical response after cessation of plasma exchange, maintained for > 30 days. The number of patients that achieved clinical remission and their frequency will be reported
TTP Exacerbation rate | Throughout the study period, approximately 3 years per patient
  Defined as a reduction in platelet count to below the lower limit of the established reference range, an increased LDH level, and the need to restart plasma exchange within 30 days of the last plasma exchange after a clinical response to plasma exchange. The number of patients with exacerbations and their frequency will be reported
TTP Relapse rate | Throughout the study period, approximately 3 years per patient
  Defined as a fall in platelet count to below the lower limit of the established reference range, with or without clinical symptoms, > 30 days after stopping of plasma exchange for an acute TTP episode, requiring reinitiation of therapy. This is usually associated with a new increase in the LDH level. The number of patients with relapse and their frequency will be reported.
Refractory TTP rate | Throughout the study period, approximately 3 years per patient
  defined as persistent thrombocytopenia, lack of a sustained platelet count increment or low platelet counts and a persistently raised LDH level despite five plasma exchanges 44 and steroid treatment. The number of patients with refractory TTP and their frequency will be reported.
Time-to-response (TTR) | Throughout the study period, approximately 3 years per patient
  Defined as the time from the date of first administration of treatment until the date of clinical response. Patients who die, are lost to follow-up, or reach the time point of analysis without a known record of response will have the TTR censored at the date of death, last assessment or last contact of a follow-up, whichever occurs last. Patients who received a new treatment for TTP whatever the type of treatment before disease response will be censored at the start date of this new treatment. The cumulative incidence of TTR will be estimated by the method of Kaplan-Meier.
Duration of response (DoR) | Throughout the study period, approximately 3 years per patient
  DoR will be calculated among those patients that achieve a clinical response from the time that measurement criteria are first met until the date of exacerbation, relapse, appearance of refractory TTP or death by any cause. Patients who are lost to follow-up, or reach the time point of analysis without a known record of TTP recurrence or death will have the DoR censored at the date of last assessment or last contact of a follow-up, whichever occurs last. Patients who received a new treatment for TTP, whatever the type of treatment, will be censored at the start date of this new treatment.
Relapse-free survival (RFS) | Throughout the study period, approximately 3 years per patient
  RFS will be calculated from the date of first administration of treatment until the date of TTP relapse or the date of death due to any cause. Patients who are lost to follow-up, or reach the time point of analysis without a known record of relapse or death will have the RFS censored at the date of last assessment or last contact, whichever occurs last. Patients who received a new treatment for TTP, whatever the type of treatment, before disease relapse or death will be censored at the start date of this new treatment. The cumulative incidence of relapse will be estimated by the method of Kaplan-Meier
Overall survival (OS) | Throughout the study period, approximately 3 years per patient
  OS will be calculated from the date of the first episode recorded until the date of death due to any cause. Patients who are lost to follow-up or reach the time point of analysis without a known record of death will have the OS censored at the date of last contact. The cumulative incidence of OS will be estimated by the method of Kaplan-Meier.
Frequency of serious adverse events (SAEs) | Throughout the study period, approximately 3 years per patient
  Percentage of patients who experience SAEs during the study
Rate of complications associated with plasma exchange treatment | Throughout the study period, approximately 3 years per patient
  Percentage of patients who experience complications associated with plasma exchange
Frequency of complications associated with plasma exchange treatment | Throughout the study period, approximately 3 years per patient
  Number of complications associated with plasma exchange per TTP event

CONTACTS AND LOCATIONS:
Overall Officials: Dr. María Eva Mingot Castellano, M.D. Ph.D., Study Chair — Hospital Universitario Virgen del Rocío. Sevilla, España.
Locations (7):
- Spain (7):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Universitario Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínic Barcelona, Barcelona
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitario La Paz, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided